CLINICAL TRIAL: NCT02004119
Title: Randomized Double-blind Placebo-controlled Study of KHK4577 in Patients With Atopic Dermatitis
Brief Title: Phase 2 Study of KHK4577
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4577-002
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KHK4577 (Experimental)
  Interventions: Drug: KHK4577

INTERVENTIONS:
Drug: KHK4577
  Arms: KHK4577
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is an randomized double-blind placebo-controlled study to evaluate the efficacy and the safety of oral KHK4577 for 6 weeks in patients with atopic dermatitis. Pharmacokinetics of KHK4577 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed voluntarily the written informed consent form to participate in this study.
* Subject has been diagnosed as atopic dermatitis according to Guidelines for Management of Atopic Dermatitis (2009).
* Rajka & Langeland criteria of >/= 4.5 at screening visit
* Investigator's Global Assessment (IGA) score of >/= 3 at screening visit

Exclusion Criteria:

* Evidence of skin disorders/conditions that would interfere with the assessment of the effect of the study drug.
* Subject received photochemotherapy or systemic immunosuppressants within 2 weeks prior to informed consent.
* Subject has any active infectious disease(except localized infection) which needs to treat with systemic antibiotics(eg. antibacterial, antifungal or antiviral drugs) within 4 weeks prior to informed consent.
* Subject has complications / history of drug abuse or alcoholism.
* Subject has drug allergy or history of allergic reaction to a drug medicine.
* Subject has a significant concurrent medical conditions as defined in the study protocol.
* Subject is breast-feeding, pregnant or planning to become pregnant in this study period.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent improvement from baseline in Eczema Area and Severity Index (EASI) | Pre-dose, Week 1,2,4 and 6

SECONDARY OUTCOMES:
Change from baseline in Investigator's Global Assessment score | Pre-dose, Week 1,2,4 and 6
Dermatology Life Quality Index | Pre-dose, Week 1,2,4 and 6
Visual Analog Scale (itching) | Pre-dose, Week 1,2,4 and 6
Incidence of patients with adverse events | From Day 1 through Week 6
Profile of pharmacokinetics of plasma KHK4577 concentration | pre-dose, Week 1,2,4 and 6

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Sapporo, Hokkaido, Japan